CLINICAL TRIAL: NCT04490759
Title: Reference Range Pilot Study for the Quantra Analyzer With the QStat Cartridge
Brief Title: QStat Pilot Reference Range Study
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-020
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy volunteers: Blood samples from healthy volunteers analyzed on the Quantra System
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: QStat Cartridge

SUMMARY:
The objective is to determine the initial reference range intervals for the parameters reported by the Quantra System with the QStat Cartridge.

DETAILED DESCRIPTION:
This is a single center prospective, observational study of a healthy adult population with normal coagulation function to determine the initial reference range intervals for the parameters reported by the Quantra System with the QStat Cartridge. The threshold for the Clot Stability to Lysis (CSL) parameter will be determined from the CSL reference range.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject is willing to participate and has signed a consent form
* Subject's laboratory coagulation test results at screening are within each test's normal reference range.

Exclusion Criteria:

* Subject is younger than 18 years
* Subject has a history of a coagulation disorder
* Subject is pregnant or lactating
* Subject is currently taking medications known to alter coagulation
* Subject has one or more laboratory coagulation test restuls outside of the normal reference range at screening
* Subject had a blood transfusion or surgery within the last month
* Drug abuse
* Excessive alcohol consumption
* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers with normal coagulation function, approximately equal numbers of males and females across three age group categories (18-30, 31-50 and >50 years). The racial and ethnic profiles will be representative of the populations at the site.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Reference range intervals for measurement of Clot Time (CT) parameter | Baseline, determined from a single blood draw
  Reference range intervals determined in this study will serve as the reference range for CT on the QStat Cartridge when it is commercially available.
Reference range intervals for measurement of Clot Stiffness (CS) parameter | Baseline, determined from a single blood draw
  Reference range intervals determined in this study will serve as the reference range for CS on the QStat Cartridge when it is commercially available.
Reference range intervals for measurement of Fibrinogen Contribution to Clot Stiffness (FCS) parameter | Baseline, determined from a single blood draw
  Reference range intervals determined in this study will serve as the reference range for FCS on the QStat Cartridge when it is commercially available.
Reference range intervals for measurement of Platelet Contribution to Clot Stiffness (PCS) parameter | Baseline, determined from a single blood draw
  Reference range intervals determined in this study will serve as the reference range for PCS on the QStat Cartridge when it is commercially available.
Reference range intervals for measurement of Clot Stability to Lysis (CSL) parameter | Baseline, determined from a single blood draw
  Reference range intervals determined in this study will serve as the reference range for CSL on the QStat Cartridge when it is commercially available.

CONTACTS AND LOCATIONS:
Locations (1):
- M3 Wake Research, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No